CLINICAL TRIAL: NCT06353932
Title: The Effect of Monitoring Endotracheal Tube Cuff Pressure and Keeping it in a Certain Range on the Incidence of Post-surgery Cough, Sore Throat, Hoarseness.
Brief Title: The Effect of Monitoring Endotracheal Tube Cuff Pressure and Keeping it in a Certain Range
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kheyrana Mahmudova, Principal İnvestigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KA-23026
Record Dates: First submitted 2024-03-14; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Endotracheal Tube; Cuff Pressure; Sore Throat
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The endotracheal tubes of the control group were placed and inflated by the caregiver. A seperate blinded researcher measured cuff pressures by manometer but did not inform the team and no intervention was made.
- study group (Active Comparator): The endotracheal tube cuff pressures of the study group patients were constantly monitored and kept within the range of 20-25 cm H2O.
  Interventions: Other: keeping the endotracheal tube cuff pressure within a certain range

INTERVENTIONS:
Other: keeping the endotracheal tube cuff pressure within a certain range — The endotracheal tube cuff pressures of the study group patients were kept within the range of 20-25 cm H2O.
  Other Names: measuring ETT cuff pressures with a manometer and continuous pressure monitor
  Arms: study group

SUMMARY:
The main purpose of our prospective, randomized, controlled, double-blind study is to investigate the effect of keeping endotracheal tube cuff pressures within a certain range on the incidence of postoperative sore throat, hoarseness and cough.The secondary aims of our study are to evaluate the effect of intubation duration, smoking, presence of chest disease, presence of blood on the intubation tube after extubation, presence of NG\OG, and type of surgery on the incidence of sore throat, hoarseness, and cough.The patients were randomly divided into two: a study group with continuous cuff pressure monitoring and a control group without continuous cuff pressure monitoring.The endotracheal cuff pressure of the patients in both groups was measured by a blinded researcher using a cuff manometer after intubation, before extubation, and in long cases, at the 3rd hour after intubation.Patients were evaluated for sore throat, cough, and hoarseness at the 2nd and 24th hours by another researcher blinded to the study groups.

DETAILED DESCRIPTION:
Although the safe cuff pressure range for high volume-low pressure tubes used today is defined as 20-30 cmH2O, routine cuff pressure monitoring is not performed in operating rooms. The aim of this study is to investigate whether there is a significant pressure difference between blindly inflated cuffs and the cuffs inflated by controlling the cuff pressure aided by monitorization, and the effects of any detected pressure difference on the trachea using the clinically detectable parameters of sore throat, hoarseness and cough. The patients included in this prospective, controlled, randomized, double-blind study were divided into two groups: the study group whose cuff pressures were monitored continously (n = 163) and the control group (n = 100). The study group was constantly monitored with an invasive pressure monitoring system. In addition, a researcher who was blind to the groups measured the endotracheal tube cuff pressure with the help of a manometer after intubation in both groups, before extubation, and in long-term cases, at the 3rd hour after intubation. Postoperatively, patients were evaluated for sore throat, cough, and hoarseness using VAS scoring at the 2nd and 24th hour by another researcher blinded to the study groups. Statistical evaluation was made using the Statistical Package for Social Sciences for Windows 20 (SPSS-IBM SPSS Inc., Chicago, IL) program. Complaint of sore throat was observed significantly less at 2nd and 24th hours in the group with cuff pressure monitoring (p=0.00 for 2nd hour sore throat, p=0.02 for 24th hour sore throat). No difference was detected between the groups in terms of hoarseness and cough. It has been observed that manometer measurements also reduce the pressure due to the use of air in the same closed system. The quantity of this reduction, which some researchers have previously stated, needs to be studied in more detail. In conclusion, intraoperative ETT cuff pressure monitoring may be effective in preventing sore throat and the mucosal ischemia that causes this pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA ( american society of anesthesiologists) I-II-III group patients
* elective surgery
* surgery under general anesthesia
* gynecology and obstetrics and general surgery

Exclusion Criteria:

* Patients who did not agree to participate in the study,
* Patients under 18 years of age,
* Patients with ASA IV, V, VI,
* Patients scheduled for emergency surgery,
* Patients for whom difficult intubation is anticipated
* Patients who could not be intubated on the first try.
* Patients with tracheostomy
* Thyroidectomy operations
* Parathyroidectomy operations
* COPD (Chronic Obstructive Pulmonary Disease) patients who have had an attack in the last 6 months
* Patients who complain of sore throat, hoarseness and cough before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Sore throat | second and 24th hours postoperatively
  Blinded researcher using VAS (The Visual Analogue Scale) score to evaluate patient discomfort level.0-no pain, score <3 mild pain, 3-6 moderate pain, and >6 severe pain
cough | second and 24th hours postoperatively
  Blinded researcher using yes/no to evaluate patient discomfort. yes means the patient has a cough, no means she/he does not
hoarseness | second and 24th hours postoperatively
  Blinded researcher using yes/no to evaluate patient discomfort. yes means the patient has hoarseness, no means she/he does not

CONTACTS AND LOCATIONS:
Overall Officials: Murat İzgi, Ass. Prof., Principal Investigator — Hacettepe University Department of Anesthesiology
Locations (1):
- Hacettepe University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All checked supporting information is available, stored by the investigators. If
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All data will be kept for a year after the completion of the study

REFERENCES:
- [Result] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989
- [Result] Asai S, Motoyama A, Matsumoto Y, Konami H, Imanaka H, Nishimura M. Decrease in cuff pressure during the measurement procedure: an experimental study. J Intensive Care. 2014 Jun 2;2(1):34. doi: 10.1186/2052-0492-2-34. eCollection 2014. PMID 25908987
- [Result] Liu J, Zhang X, Gong W, Li S, Wang F, Fu S, Zhang M, Hang Y. Correlations between controlled endotracheal tube cuff pressure and postprocedural complications: a multicenter study. Anesth Analg. 2010 Nov;111(5):1133-7. doi: 10.1213/ANE.0b013e3181f2ecc7. Epub 2010 Aug 24. PMID 20736432
- [Result] Yildirim ZB, Uzunkoy A, Cigdem A, Ganidagli S, Ozgonul A. Changes in cuff pressure of endotracheal tube during laparoscopic and open abdominal surgery. Surg Endosc. 2012 Feb;26(2):398-401. doi: 10.1007/s00464-011-1886-8. Epub 2011 Sep 10. PMID 21909860